CLINICAL TRIAL: NCT06132308
Title: Evaluation of PENG Block Applied in Hip Surgery in Terms of Block Duration and Postoperative Pain
Brief Title: Evaluation of PENG Block in Terms of Block Time and Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savas Altinsoy, Assistant Professor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Diskapı-YB-SA-PENG
Record Dates: First submitted 2023-03-17; First posted 2023-11-15 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain
Keywords: PENG; Hip fracture
MeSH Terms: conditions — Pain, Postoperative; Hip Fractures | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PENG Block with 0.25% bupivacaine (20 cc) (Active Comparator): For PENG block, patients are in the supine position is deposited. The convex ultrasound probe is initially placed over the anterior superior iliac spine, then the probe moves medially until the femoral artery is visualized. In this view, iliopectineal eminence (IPE), iliopsoas muscle and tendon, femoral artery and iliac muscle are observed. Between the psoas tendon and the IPE 22 gauge 80 mm block needle is guided and 20cc local anesthetic used in % 0.25 bupivacaine is administered by intermittent aspiration.
  Interventions: Procedure: PENG Block with 0.25% bupivacaine
- PENG Block with 0.25% bupivacaine (30 cc) (Experimental): For PENG block, patients are in the supine position is deposited. The convex ultrasound probe is initially placed over the anterior superior iliac spine, then the probe moves medially until the femoral artery is visualized. In this view, iliopectineal eminence (IPE), iliopsoas muscle and tendon, femoral artery and iliac muscle are observed. Between the psoas tendon and the IPE 22 gauge 80 mm block needle is guided and 30cc local anesthetic used in % 0.25 bupivacaine is administered by intermittent aspiration.
  Interventions: Procedure: PENG Block with 0.25% bupivacaine
- PENG Block with 0.25% bupivacaine (40 cc) (Experimental): For PENG block, patients are in the supine position is deposited. The convex ultrasound probe is initially placed over the anterior superior iliac spine, then the probe moves medially until the femoral artery is visualized. In this view, iliopectineal eminence (IPE), iliopsoas muscle and tendon, femoral artery and iliac muscle are observed. Between the psoas tendon and the IPE 22 gauge 80 mm block needle is guided and 40cc local anesthetic used in % 0.25 bupivacaine is administered by intermittent aspiration.
  Interventions: Procedure: PENG Block with 0.25% bupivacaine

INTERVENTIONS:
Procedure: PENG Block with 0.25% bupivacaine — Peng block was performed.

SUMMARY:
Hip fracture is a common orthopedic emergency in the elderly and causes significant morbidity and is associated with mortality. In most patients, surgical reduction and fixation is the definitive treatment. Effective perioperative analgesia minimizing the need for opioids and related side effects is recommended in this patient population. Therefore, various methods are used. When the investigators look at the literature, for PENG block It is observed that different drug doses (20cc, 30cc, and 40cc) are used. In this study, the investigators planned to investigate the effectiveness of PENG blocks, postoperative analgesia, and side effects.

DETAILED DESCRIPTION:
Patients in the ASA 1-3 group who had hip surgery with PENG block for any reason will be included in the study. Approximately 60 patients will participate in the study, the number will be finalized as a result of power analysis. The routine algorithm for patients who will undergo hip surgery is spinal or general anesthesia after peripheral block for postoperative analgesia. Before the block, all patients were monitored by standard monitoring and intravenous vascular access was opened. For PENG block, patients are in the supine position is deposited. The convex ultrasound probe is initially placed over the anterior superior iliac spine, then the probe moves medially until the femoral artery is visualized. In this view, iliopectineal eminence (IPE), iliopsoas muscle and tendon, femoral artery and iliac muscle are observed. Between the psoas tendon and the IPE 22 gauge 80 mm block needle is guided and local anesthetic is administered by intermittent aspiration. Although drug doses vary according to the patient and the surgery to be performed in our clinic, %0.25 bupivacaine is used in 20cc, 30cc and 40cc doses. In all patients with block, 30 minutes after the block application, motor and sensory examination is carried out. Sensory block was evaluated by cold stimulus (0 = no cold sensation, 1 = cold sensation severely reduced, 2 = cold sensation slightly decreased, 3 = normal cold sensation). In patients who will undergo hip surgery, due to limited kidney and liver reserves opioids are often used for analgesia. In our clinic, to reduce opioid use in this elderly patient group, preoperative nerve block method is used. Postoperative analgesic needs of the patients will be recorded from the information in the current patient controlled analgesia device. Demographic data of patients, surgical method and duration from the anesthesia form will be followed. Postoperative numerical evaluation scale (NRS-numeric rating scale; 0 = no pain, 10 = excruciating pain) will be recorded. Postoperative pain, muscle strength, block time and nausea-vomiting PACU, 4, 8, 24 hours will be recorded. Postoperative pain treatment satisfaction of patients numerically scale (NRS, 0 = dissatisfied, 10 = extremely satisfied) and postoperative first night sleep quality at 24 hours with NRS (0= could not sleep all night, 10= slept very well) query will be recorded.

ELIGIBILITY:
Inclusion Criteria:

- Patients who have undergone hip surgery with PENG block for any reason

Exclusion Criteria:

* chronic opioid users
* cognitive disorders
* written consent form haven't get
* history of relevant drug allergy
* infection of the skin at the site of needle puncture area
* coagulopathy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
The degree of postoperative pain | 0 hour
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
The degree of postoperative pain | 4 hour
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
The degree of postoperative pain | 8 hour
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
The degree of postoperative pain | 24 hour
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
Postoperative tramadol consumption | 24 hour
  total tramadol consumption in three groups will be assessed in the postoperative period

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Department of Anesthesiology and Reanimation, University of Health Sciences, Diskapi Yıldırım Beyazit Training and Research Hospital, Ankara
  - university of health siences diskapi yildirim beyazit T&R hospital, Ankara

IPD SHARING:
Plan to Share IPD: No